CLINICAL TRIAL: NCT06246747
Title: The Use of Telerehabilitation to Improve Movement-related Outcomes and Quality of Life for Patients With Parkinson's Disease: A Pilot Randomized Controlled Trial
Brief Title: The Use of Telerehabilitation to Improve Movement Outcomes for Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wizecare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00005367
Record Dates: First submitted 2023-12-14; First posted 2024-02-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; physical therapy; telerehabilitation; satisfaction; adherence to home exercise
MeSH Terms: conditions — Parkinson Disease; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical therapy treatment in the clinic + telerehabilitation (Experimental): Patients performed treatments in the clinic in the presence of their physical therapist (PT) as well as perform remote treatment from their homes. The remote treatment included using video chat with their PT as well as performing PD-specific exercises which were stored in a specific library on the platform.
  Interventions: Other: In clinic physical therapy; Other: Telerehabilitation only
- TR-only (Experimental): Patients received treatment at their homes using the TR platform. This included video chat with their clinician as well as performing PD-specific exercises which were stored in a specific library on the platform.
  Interventions: Other: Telerehabilitation only
- Control group (Active Comparator): Patients received treatment in the clinic in the presence of their PT
  Interventions: Other: In clinic physical therapy

INTERVENTIONS:
Other: In clinic physical therapy — Patients visit the clinic to receive traditional physical therapy treatment
  Arms: Control group; Physical therapy treatment in the clinic + telerehabilitation
Other: Telerehabilitation only — Patients receive remote treatment using the Wizecare platform
  Other Names: Wizecare Telerehabilitation Platform
  Arms: Physical therapy treatment in the clinic + telerehabilitation; TR-only

SUMMARY:
The goal of this pilot randomized clinical trial was to assess the feasibility of telerehabilitation (TR) for patients with Parkinson&amp;#39;s Disease (PD). The main questions it aims to answer are: 1. whether the recruitment to such a study will be successful and the satisfaction of both participants and clinicians will be good. 2. Clinical effectiveness of TR for patients with PD was also explored. Participants were randomized to 3 groups : 1. Clinic+TR. 2. TR-only group and 3. A usual control group. Results were compared between the groups.

DETAILED DESCRIPTION:
Patients were identified for pre-screening if they had a diagnosis of PD for any duration and were scheduled for a new episode of physical therapy. Pre-screening included chart review by a study coordinator. The exclusion criteria were: any outpatient physical therapy episode in the preceding 5 months, documented diagnosis of another progressive neurological disease, history of epilepsy, moderate to severe cognitive impairment, hemiparesis or hemiplegia, current complaints of dizziness. Though not an a priori criterion, some patients could not be scheduled for study participation due to a lack of availability on the schedules of participating therapists.

Those meeting eligibility criteria were contacted in writing (via mailed letter or electronic health record portal) then via phone by a coordinator two to four weeks prior to their initial physical therapy visit. At pre-screen phone call, patients were excluded if they were not reached, reported not having a reliable caregiver or internet connection in their home, or declined to participate.

After chart review and phone screening, those interested in participation were consented in-person by the study coordinator and further screened for eligibility by the evaluating physical therapist immediately prior to their initial physical therapy visit. Final eligibility was determined by completion of the timed-up-and-go test (TUG) less than15 seconds, a 10-meter gait speed of more than 0.8 m/s, and a subjective determination of safety by the evaluating physical therapist.

The primary intervention of interest in this study was the delivery of physical therapist interventions using a TR platform (WizeCare Technologies, Or Yehuda, Israel). Patients completed TR on a tablet (Lenovo Yoga Tab 3, Model YT3-X50F, OS Android 6.0) provided by WizeCare, their own tablet, their own laptop or desktop computer, or their own cell phone. If by tablet or cell phone, the platform was accessed using a mobile app. If by computer, the platform was accessed via the internet.

The WizeCare TR platform enables remote rehabilitation training and monitoring using a customized combination of video conferencing and libraries of pre-recorded videos of specific exercises. These videos can be combined manually to create unique exercise plans for patients that vary in content and duration. Immediately prior to this study, a series of videos of common PD-specific exercises were produced and stored in a specific library on the platform. Physical therapists built customized home exercise programs primarily from this library, though videos from any library were available for use. The platform also features an option for live video calls between patients and therapists, which enabled ongoing communication and re-evaluation for manual adjustment of the rehabilitation plan as needed.

Baseline demographic variables were age and gender. Baseline clinical variables were years since PD diagnosis, the modified Hoehn and Yahr scale, and the Unified Parkinson's Disease Rating Scale (UPDRS). Hoehn and Yahr stages range from 1 (unilateral involvement only) to 5 (wheelchair-bound or bedridden unless aided), with the modified scale including stages 1.5 and 2.5 to account for intermediate phases of disease progression. The UPDRS is a clinician-rated instrument of observable PD symptoms that are assessed for four different constructs: mental dysfunction and mood, activities of daily living, motor function, and treatment-related complications; higher UPDRS total scores indicate greater symptom severity.

At each interaction with the treating physical therapist-in clinic or via the TR platform-subjective feedback was provided verbally by the patient regarding the safety of the exercises he or she completed at home. This is consistent with current standard practice. Any reported fall or other adverse event, whether in conjunction with the exercise program or otherwise, was reviewed by the study team (the four treating physical therapists and the PI). These were recorded and reported to the Institutional Review Board as required.

Additionally, the WizeCare platform enables a safety assessment with each session in which a patient interacts with the system, including their unsupervised home exercise sessions. At the conclusion of each session on the platform, patients are asked, "Did the patient feel safe during this session?" If they answer "No", the system can send an automated message to the treating physical therapist. The system also provides an automated response to the patient to, "Please stop participating in the exercise program and call the treating physical therapist." Initiated by either the physical therapist or the patient within 24 hours of the reported lack of safety, a conversation between them will allow the patient to express their safety concerns. Any such events were recorded as adverse events, with subsequent steps as outlined above. These patient self-reports of safety were included amongst exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 with PD of any duration
* The patient was scheduled for a new episode of physical therapy.

Exclusion Criteria:

* Any outpatient physical therapy episode in the preceding 5 months
* Documented diagnosis of another progressive neurological disease
* History of epilepsy
* Moderate to severe cognitive impairment
* Hemiparesis or hemiplegia
* Current complaints of dizziness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Satisfaction assessment | From enrollment to end of treatment at 5 weeks
  We assessed satisfaction with the mode of care delivery using novel surveys, which were administered to the patient and the physical therapist at the in-clinic discharge visit via the Research Electronic Data Captureapture (REDCap) platform. Each survey assessed eight constructs; six satisfaction items were rated on a 5-point Likert scale ("very poor", "poor", "fair", "good", or "very good"). The number 1 stood for "very poor" and the number 5 stood for "very good". The item pertaining to safety asked for a 0 ("very unsafe") to 100 ("very safe") rating.

SECONDARY OUTCOMES:
Clinical effectiveness of TR | From enrollment to end of treatment at 5 weeks
  Clinical effectiveness was measured by the Parkinson's Disease Questionnaire (PDQ-39) which is a self-reported questionnaire. It consists of 39 items across eight domains: Mobility, Activities of Daily Living, Emotional Well-being, Stigma, Social Support, Cognition, Communication, and Bodily Discomfort. Each item is rated on a scale from 0 to 4, with 0 representing no difficulty and 4 representing severe difficulty. Scores are calculated by summing the responses for each domain and transforming them into a score ranging from 0 to 100, with higher scores indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stilphen, PT, DPT, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleavelnad Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds GO, Otto MW, Ellis TD, Cronin-Golomb A. The Therapeutic Potential of Exercise to Improve Mood, Cognition, and Sleep in Parkinson's Disease. Mov Disord. 2016 Jan;31(1):23-38. doi: 10.1002/mds.26484. Epub 2015 Dec 30. PMID 26715466
- [Background] van der Kolk NM, King LA. Effects of exercise on mobility in people with Parkinson's disease. Mov Disord. 2013 Sep 15;28(11):1587-96. doi: 10.1002/mds.25658. PMID 24132847
- [Background] Goodwin VA, Richards SH, Taylor RS, Taylor AH, Campbell JL. The effectiveness of exercise interventions for people with Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2008 Apr 15;23(5):631-40. doi: 10.1002/mds.21922. PMID 18181210
- [Background] Corcos DM, Robichaud JA, David FJ, Leurgans SE, Vaillancourt DE, Poon C, Rafferty MR, Kohrt WM, Comella CL. A two-year randomized controlled trial of progressive resistance exercise for Parkinson's disease. Mov Disord. 2013 Aug;28(9):1230-40. doi: 10.1002/mds.25380. Epub 2013 Mar 27. PMID 23536417
- [Background] Shulman LM, Katzel LI, Ivey FM, Sorkin JD, Favors K, Anderson KE, Smith BA, Reich SG, Weiner WJ, Macko RF. Randomized clinical trial of 3 types of physical exercise for patients with Parkinson disease. JAMA Neurol. 2013 Feb;70(2):183-90. doi: 10.1001/jamaneurol.2013.646. PMID 23128427
- [Background] Wu PL, Lee M, Huang TT. Effectiveness of physical activity on patients with depression and Parkinson's disease: A systematic review. PLoS One. 2017 Jul 27;12(7):e0181515. doi: 10.1371/journal.pone.0181515. eCollection 2017. PMID 28749970
- [Background] Ahlskog JE. Does vigorous exercise have a neuroprotective effect in Parkinson disease? Neurology. 2011 Jul 19;77(3):288-94. doi: 10.1212/WNL.0b013e318225ab66. PMID 21768599
- [Background] King LA, Wilhelm J, Chen Y, Blehm R, Nutt J, Chen Z, Serdar A, Horak FB. Effects of Group, Individual, and Home Exercise in Persons With Parkinson Disease: A Randomized Clinical Trial. J Neurol Phys Ther. 2015 Oct;39(4):204-12. doi: 10.1097/NPT.0000000000000101. PMID 26308937
- [Background] Ferraz DD, Trippo KV, Duarte GP, Neto MG, Bernardes Santos KO, Filho JO. The Effects of Functional Training, Bicycle Exercise, and Exergaming on Walking Capacity of Elderly Patients With Parkinson Disease: A Pilot Randomized Controlled Single-blinded Trial. Arch Phys Med Rehabil. 2018 May;99(5):826-833. doi: 10.1016/j.apmr.2017.12.014. Epub 2018 Jan 11. PMID 29337023
- [Background] Qiang JK, Marras C. Telemedicine in Parkinson's disease: A patient perspective at a tertiary care centre. Parkinsonism Relat Disord. 2015 May;21(5):525-8. doi: 10.1016/j.parkreldis.2015.02.018. Epub 2015 Feb 28. PMID 25791380
- [Background] Wilkinson JR, Spindler M, Wood SM, Marcus SC, Weintraub D, Morley JF, Stineman MG, Duda JE. High patient satisfaction with telehealth in Parkinson disease: A randomized controlled study. Neurol Clin Pract. 2016 Jun;6(3):241-251. doi: 10.1212/CPJ.0000000000000252. PMID 27347441
- [Background] Dorsey ER, Vlaanderen FP, Engelen LJ, Kieburtz K, Zhu W, Biglan KM, Faber MJ, Bloem BR. Moving Parkinson care to the home. Mov Disord. 2016 Sep;31(9):1258-62. doi: 10.1002/mds.26744. Epub 2016 Aug 8. PMID 27501323
- [Background] Fullard ME, Thibault DP, Hill A, Fox J, Bhatti DE, Burack MA, Dahodwala N, Haberfeld E, Kern DS, Klepitskava OS, Urrea-Mendoza E, Myers P, Nutt J, Rafferty MR, Schwalb JM, Shulman LM, Willis AW; Parkinson Study Group Healthcare Outcomes and Disparities Working Group. Utilization of rehabilitation therapy services in Parkinson disease in the United States. Neurology. 2017 Sep 12;89(11):1162-1169. doi: 10.1212/WNL.0000000000004355. Epub 2017 Aug 23. PMID 28835397
- [Background] Prvu Bettger J, Resnik LJ. Telerehabilitation in the Age of COVID-19: An Opportunity for Learning Health System Research. Phys Ther. 2020 Oct 30;100(11):1913-1916. doi: 10.1093/ptj/pzaa151. No abstract available. PMID 32814976
- [Background] Middleton A, Simpson KN, Bettger JP, Bowden MG. COVID-19 Pandemic and Beyond: Considerations and Costs of Telehealth Exercise Programs for Older Adults With Functional Impairments Living at Home-Lessons Learned From a Pilot Case Study. Phys Ther. 2020 Aug 12;100(8):1278-1288. doi: 10.1093/ptj/pzaa089. PMID 32372072
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Poewe W. Clinical measures of progression in Parkinson's disease. Mov Disord. 2009;24 Suppl 2:S671-6. doi: 10.1002/mds.22600. PMID 19877235
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Brusse KJ, Zimdars S, Zalewski KR, Steffen TM. Testing functional performance in people with Parkinson disease. Phys Ther. 2005 Feb;85(2):134-41. PMID 15679464
- [Background] Dal Bello-Haas V, Klassen L, Sheppard MS, Metcalfe A. Psychometric Properties of Activity, Self-Efficacy, and Quality-of-Life Measures in Individuals with Parkinson Disease. Physiother Can. 2011 Winter;63(1):47-57. doi: 10.3138/ptc.2009-08. Epub 2011 Jan 20. PMID 22210979
- [Background] Cekok K, Kahraman T, Duran G, Donmez Colakoglu B, Yener G, Yerlikaya D, Genc A. Timed Up and Go Test With a Cognitive Task: Correlations With Neuropsychological Measures in People With Parkinson's Disease. Cureus. 2020 Sep 22;12(9):e10604. doi: 10.7759/cureus.10604. PMID 33123423
- [Background] Duncan RP, Leddy AL, Earhart GM. Five times sit-to-stand test performance in Parkinson's disease. Arch Phys Med Rehabil. 2011 Sep;92(9):1431-6. doi: 10.1016/j.apmr.2011.04.008. PMID 21878213
- [Background] Paul SS, Canning CG, Sherrington C, Fung VS. Reproducibility of measures of leg muscle power, leg muscle strength, postural sway and mobility in people with Parkinson's disease. Gait Posture. 2012 Jul;36(3):639-42. doi: 10.1016/j.gaitpost.2012.04.013. Epub 2012 May 27. PMID 22640867
- [Background] Steffen T, Seney M. Test-retest reliability and minimal detectable change on balance and ambulation tests, the 36-item short-form health survey, and the unified Parkinson disease rating scale in people with parkinsonism. Phys Ther. 2008 Jun;88(6):733-46. doi: 10.2522/ptj.20070214. Epub 2008 Mar 20. Erratum In: Phys Ther. 2010 Mar;90(3):462. PMID 18356292
- [Background] Leddy AL, Crowner BE, Earhart GM. Utility of the Mini-BESTest, BESTest, and BESTest sections for balance assessments in individuals with Parkinson disease. J Neurol Phys Ther. 2011 Jun;35(2):90-7. doi: 10.1097/NPT.0b013e31821a620c. PMID 21934364
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Stiggelbout AM, Van der Weijden T, De Wit MP, Frosch D, Legare F, Montori VM, Trevena L, Elwyn G. Shared decision making: really putting patients at the centre of healthcare. BMJ. 2012 Jan 27;344:e256. doi: 10.1136/bmj.e256. PMID 22286508
- [Background] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Background] Cottrell MA, Galea OA, O'Leary SP, Hill AJ, Russell TG. Real-time telerehabilitation for the treatment of musculoskeletal conditions is effective and comparable to standard practice: a systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):625-638. doi: 10.1177/0269215516645148. Epub 2016 May 2. PMID 27141087
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Flynn A, Preston E, Dennis S, Canning CG, Allen NE. Home-based exercise monitored with telehealth is feasible and acceptable compared to centre-based exercise in Parkinson's disease: A randomised pilot study. Clin Rehabil. 2021 May;35(5):728-739. doi: 10.1177/0269215520976265. Epub 2020 Dec 3. PMID 33272025
- [Background] Quinn L, Macpherson C, Long K, Shah H. Promoting Physical Activity via Telehealth in People With Parkinson Disease: The Path Forward After the COVID-19 Pandemic? Phys Ther. 2020 Sep 28;100(10):1730-1736. doi: 10.1093/ptj/pzaa128. PMID 32734298
- [Background] van den Bergh R, Evers LJW, de Vries NM, Silva de Lima AL, Bloem BR, Valenti G, Meinders MJ. Usability and utility of a remote monitoring system to support physiotherapy for people with Parkinson's disease. Front Neurol. 2023 Oct 12;14:1251395. doi: 10.3389/fneur.2023.1251395. eCollection 2023. PMID 37900610
- [Background] Cornforth E. Telerehabilitation Has Potential, But More Research, Funding, And Advocacy Are Needed. Health Affairs Forefront. Published online January 5, 2023
- [Background] Chatto CA, York PT, Slade CP, Hasson SM. Use of a Telehealth System to Enhance a Home Exercise Program for a Person With Parkinson Disease: A Case Report. J Neurol Phys Ther. 2018 Jan;42(1):22-29. doi: 10.1097/NPT.0000000000000209. PMID 29206708
- [Background] Barksdale H, McHugh B, Hodges W, Peters J, Smotherman C, Hoffman PM. Tele-Rehabilitation for Individuals with Multiple Sclerosis and Mobility Disorders-A Feasibility and Pilot Study. Telehealth and Medicine Today. 2020;5(4).
- [Derived] Johnson JK, Longhurst JK, Gevertzman M, Jefferson C, Linder SM, Bethoux F, Stilphen M. The Use of Telerehabilitation to Improve Movement-Related Outcomes and Quality of Life for Individuals With Parkinson Disease: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Jul 31;8:e54599. doi: 10.2196/54599. PMID 39083792
- Available data/document: Study Protocol — https://drive.google.com/file/d/1F2ZuHApDf800Q9Tox-sujdf0sHmctTO0/view?usp=sharing — The protocol can be accessed by clicking the Google Drive link above. For any additional questions or an issue with opening the link, please contact bella@wizecare.com